CLINICAL TRIAL: NCT01978093
Title: Immunogenicity, Safety and Reactogenicity of GSK Biologicals' Hib-MenCY-TT (MenHibrix®) Vaccine 792014 Compared to Merck & Co, Inc. Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) Vaccine in Healthy Infants and Toddlers
Brief Title: Immunogenicity, Safety and Reactogenicity Study of GlaxoSmithKline (GSK) Biologicals' Hib-MenCY-TT (MenHibrix®) Vaccine Compared to Merck & Co, Inc. PedvaxHIB Vaccine in Healthy Infants and Toddlers 12 to 15 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112931; 2013-003459-39 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
Keywords: Conjugate; Immunogenicity; Hib-MenCY-TT vaccine; Haemophilus type b; Safety; Reactogenicity
MeSH Terms: conditions — Haemophilus Infections | interventions — Hib-MenCY-TT vaccine; PEDIARIX; RIX4414 vaccine; 13-valent pneumococcal vaccine; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine; Hepatitis A Vaccines

ARMS (2):
- HibCY Group (Experimental): Subjects received 4 doses of Hib-MenCY-TT (MenHibrix®) vaccine at Day 0, Month 2, Month 4 and Month 10-13 , 3 doses of Pediarix® vaccine at Day 0, Month 2 and Month 4, 2 doses of Rotarix® vaccine at Day 0 and Month 2, 4 doses of Prevnar 13® vaccine at Day 0 and Month 2, Month 4 and Month 10-13 and 2 doses of Havrix® vaccine at Month 10-13 and Month 16-19.
  Interventions: Biological: Hib-MenCY-TT (MenHibrix®); Biological: Pediarix®; Biological: Rotarix®; Biological: Prevnar 13®; Biological: Havrix®
- PedHIB Group (Active Comparator): Subjects received 3 doses of PedvaxHIB® vaccine at Day 0, Month 2 and Month 10-13, 3 doses of Pediarix® vaccine at Day 0, Month 2 and Month 4, 2 doses of Rotarix® vaccine at Day 0 and Month 2, 4 doses of Prevnar 13® vaccine at Day 0 and Month 2, Month 4 and Month 10-13 and 2 doses of Havrix® vaccine at Month 10-13 and Month 16-19.
  Interventions: Biological: Pediarix®; Biological: Rotarix®; Biological: Prevnar 13®; Biological: PedvaxHIB®; Biological: Havrix®

INTERVENTIONS:
Biological: Hib-MenCY-TT (MenHibrix®) — 4 doses administered intramuscularly (IM) in the right upper anterolateral thigh at Day 0, Month 2, Month 4 and Month 10-13 in the HibCY Group.
  Arms: HibCY Group
Biological: Pediarix® — 3 doses administered IM in the left upper anterolateral thigh at Day 0, Month 2 and Month 4. 2 doses administered IM in the left upper anterolateral thigh at Day 0 and Month 2 and 1 dose administered IM in the right upper anterolateral thigh at Month 4 in the PedHIB Group.
Biological: Rotarix® — 2 doses administered orally at Day 0 and Month 2 each in the HibCY Group and PedHIB Group.
Biological: Prevnar 13® — 4 doses administered IM in the left lower anterolateral thigh at Day 0, Month 2, Month 4 and Month 10-13 each in the HibCY Group and PedHIB Group.
Biological: PedvaxHIB® — 3 doses administered IM in the right upper anterolateral thigh at Day 0, Month 2 and Month 10-13 in the PedHIB Group.
  Arms: PedHIB Group
Biological: Havrix® — 2 doses administered IM in the left upper anterolateral thigh at Month 10-13 and Month 16-19 each in the HibCY Group and PedHIB Group.

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of GSK Biologicals' Hib-MenCY-TT (MenHibrix®) vaccine co-administered with Rotarix, Prevnar 13 and Havrix as compared to PedvaxHIB co-administered with Rotarix, Prevnar 13 and Havrix in infants and toddlers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term (i.e. born after a gestation period of at least 37 weeks inclusive).
* Infants who have not received a previous dose of hepatitis B vaccine or those who have received only 1 dose of hepatitis B vaccine administered at least 30 days prior to enrollment.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth prior to the first vaccine dose. Inhaled and topical steroids are allowed.
* Previous vaccination against Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, rotavirus, pneumococcus, hepatitis A and/or poliovirus; more than one previous dose of hepatitis B vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of vaccines. Subjects may receive inactivated influenza vaccine or pandemic influenza vaccines any time during the study according to the national recommendation. Measles, mumps, rubella and varicella vaccination are allowed 30 days before or 30 days after the final vaccination of Hib-MenCY-TT or PedvaxHIB.
* History of Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, pneumococcus, hepatitis B, hepatitis A, rotavirus, and/or poliovirus disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including dry natural latex rubber. Hypersensitivity to any component of the vaccines, including gelatin or neomycin.
* Major congenital defects or serious chronic illnesses.
* History of any neurologic disorders or seizures. A single, simple febrile seizure is allowed.
* Subjects with history of intussusceptions or uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusceptions.
* Acute disease and/or fever at the time of enrollment.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2014-02-01; Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (26):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Syracuse, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 600 subjects were recruited from 27 centers in the United States. The study consists of 2 epochs: Epoch 001: starting at Day 0 and ending at the day preceding the 4th vaccination (Month 10-13) and Epoch 002: starting at Month 10-13 and ending at Month 17-20, 31 days after the 2nd Havrix vaccination
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- HibCY Group: Subjects received 4 doses of Hib-MenCY-TT vaccine at Day 0, Month 2, Month 4 and Month 10-13, 3 doses of Pediarix vaccine at Day 0, Month 2 and Month 4, 2 doses of Rotarix vaccine at Day 0 and Month 2, 4 doses of Prevnar 13 vaccine at Day 0 and Month 2, Month 4 and Month 10-13 and 2 doses of Havrix vaccine at Month 10-13 and Month 16-19.
- PedHIB Group: Subjects received 3 doses of PedvaxHIB vaccine at Day 0, Month 2 and Month 10-13, 3 doses of Pediarix vaccine at Day 0, Month 2 and Month 4, 2 doses of Rotarix vaccine at Day 0 and Month 2, 4 doses of Prevnar 13 vaccine at Day 0 and Month 2, Month 4 and Month 10-13 and 2 doses of Havrix vaccine at Month 10-13 and Month 16-19.
Period: Overall Study
Arm/Group | HibCY Group | PedHIB Group
Started | 297 | 303
Completed | 232 | 230
Not Completed | 65 | 73
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 5
Not completed — Protocol Violation | 8 | 2
Not completed — Withdrawal by Subject | 29 | 25
Not completed — Lost to Follow-up | 11 | 15
Not completed — Migrated/moved from study area | 11 | 13
Not completed — Loss of kaiser coverage | 4 | 10
Not completed — Lost kaiser health plan unable to contac | 1 | 0
Not completed — Mother lost custody of child | 0 | 1
Not completed — Child was in care of grandmother | 0 | 1
Not completed — N/A for vaccine administration | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HibCY Group | PedHIB Group | Total
Number analyzed (Participants) | 297 | 303 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 297 | 303 | 600
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (1.1) | 8.6 (1.1) | 8.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 140 | 288
  Male | 149 | 163 | 312
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 29 | 19 | 48
  American Indian or Alaskan Native | 11 | 12 | 23
  Asian - Central/South Asian Heritage | 5 | 4 | 9
  Asian - East Asian Heritage | 2 | 2 | 4
  Asian - Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 6 | 8
  White - Arabic / North African Heritage | 1 | 2 | 3
  White - Caucasian / European Heritage | 201 | 218 | 419
  Unspecified | 36 | 32 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Anti-Polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations Greater Than or Equal to (≥) 1.0 µg/mL
Description: Percentage of subjects with Anti-PRP antibody concentrations≥1.0 µg/mL were assessed.
  Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts. Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.As per an hierarchical procedure, the primary objective about Anti-PRP will first need to be met to be able to conclude on any other primary objective, and within each subsequent arm, the first primary objective will have to be reached to conclude on the second primary objective of that Epoch.
Time Frame: 1 month after the fourth dose for HibCY Group and 1 month after third dose for PedHIB Group [Month (M) 11-14]
Population: The analysis was performed on the Fourth dose According to Protocol (ATP) cohort for analysis of immunogenicity, which included all evaluable subjects who have received 3 vaccine doses in the first 3-doses vaccination course and who have received the fourth vaccine dose and the first Havrix dose.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 223 | 218
Percentage of subjects | 98.2 [95.5 to 99.5] | 97.2 [94.1 to 99.0]
Statistical Analysis 1: Comparison: HibCY Group vs PedHIB Group; Difference between HibCY and PedHIB groups in percentage of subjects with anti-PRP concentrations equal to or above the cut-off value of 1.0 µg/mL one month after the fourth dose in HibCY Group and third dose in PedHIB Group; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% CI for the difference (HibCY group minus the PedHIB group) in the percentage of subjects with anti-PRP concentrations ≥1.0 mg/mL is to be≥-10% (clinical limit for non-inferiority); Group difference in proportions; Before concluding on the primary objectives for Rotarix, Prevnar 13 and Havrix, this primary objective regarding anti-PRP needs to be reached; Difference in percentage of subjects = 0.96, 95% CI 2-sided [-2.12 to 4.30]

2. Primary Outcome: Anti-rotavirus Serum Immunoglobulin A (IgA) Geometric Mean Concentrations (GMCs).
Description: Anti-rotavirus serum IgA was assessed by ELISA, tabulated as GMCs and expressed in Units per mililiter (U/mL).Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.
  Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.As per a hierarchical procedure, the primary objective about Anti-PRP will first need to be met to be able to conclude on any other primary objective, and within each subsequent arm, the first primary objective will have to be reached to conclude on the second primary objective of that Epoch
Time Frame: 2 months post-dose 2 of Rotarix (Month 4)
Population: The analysis was performed on the Rota ATP cohort for analysis of immunogenicity, which included all evaluable subjects who received the two doses of Rotarix vaccine and for whom immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 155 | 161
U/mL | 138.9 [104.0 to 185.5] | 115.0 [87.5 to 151.0]
Statistical Analysis 1: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for anti-Rota IgA concentrations 2 months after the second dose of Rotarix vaccine; Test type: Non-Inferiority — Non-inferiority is concluded if lower limit of the two-sided standardized asymptotic 97.5% CI on the ratio of anti-rotavirus IgA GMC (HibCY group over PedHIB group) is to be ≥0.5; ANCOVA; GMC adjusted for BS sub-cohorts;97.5% confidence interval calculated for adjusted GMC ratio(Ancova model:adjustment for BS subcohorts-pooled variance); Adjusted GMC ratios = 1.21, 97.5% CI 2-sided [0.77 to 1.90] — To be able to conclude independently on primary objectives of Epoch 001(Rotarix & Prevnar13 Post dose 3)& Epoch 002 (Havrix & Prevnar13 post dose 4),a Bonferroni correction is used in order to test these objectives(1.25% 1sided for Epoch 001 & 002)

3. Primary Outcome: Anti-Streptococcus (S) Pneumoniae GMCs
Description: Antibody concentrations against S. pneumoniae serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F were assessed by ELISA, tabulated as GMCs and expressed in µg/mL.
  Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.As per an hierarchical procedure, the primary objective about Anti-PRP will first need to be met to be able to conclude on any other primary objective, and within each subsequent arm, the first primary objective will have to be reached to conclude on the second primary objective of that Epoch.
Time Frame: 1 month post-dose 3 of Prevnar 13 (Month 5)
Population: The analysis was performed on the First three doses ATP cohort for analysis of immunogenicity, which included all evaluable subjects who have received three doses of Prevnar 13 vaccine and for whom immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- HibCY Group: Subjects received 4 doses of Hib-MenCY-TT vaccine at Day 0, Month 2, Month 4 and Month 10-13 , 3 doses of Pediarix vaccine at Day 0, Month 2 and Month 4, 2 doses of Rotarix vaccine at Day 0 and Month 2, 4 doses of Prevnar 13 vaccine at Day 0 and Month 2, Month 4 and Month 10-13 and 2 doses of Havrix vaccine at Month 10-13 and Month 16-19.
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 156 | 158
µg/mL
  Anti-1 antibody | 1.49 [1.30 to 1.70] | 1.26 [1.10 to 1.44]
  Anti-3 antibody: number analyzed (Participants) | 149 | 150
  Anti-3 antibody | 0.55 [0.48 to 0.63] | 0.48 [0.42 to 0.55]
  Anti-4 antibody | 0.81 [0.72 to 0.90] | 0.74 [0.66 to 0.84]
  Anti-5 antibody | 0.80 [0.71 to 0.91] | 0.68 [0.59 to 0.78]
  Anti-6A antibody | 1.76 [1.55 to 2.00] | 1.37 [1.18 to 1.60]
  Anti-6B antibody: number analyzed (Participants) | 154 | 158
  Anti-6B antibody | 1.00 [0.85 to 1.18] | 0.87 [0.73 to 1.05]
  Anti-7F antibody | 2.59 [2.29 to 2.93] | 2.36 [2.10 to 2.65]
  Anti-9V antibody: number analyzed (Participants) | 156 | 157
  Anti-9V antibody | 0.78 [0.69 to 0.89] | 0.63 [0.55 to 0.73]
  Anti-14 antibody: number analyzed (Participants) | 156 | 156
  Anti-14 antibody | 4.77 [4.13 to 5.52] | 4.16 [3.50 to 4.94]
  Anti-18C antibody | 0.91 [0.81 to 1.03] | 0.74 [0.65 to 0.84]
  Anti-19A antibody | 1.31 [1.17 to 1.48] | 1.13 [0.98 to 1.31]
  Anti-19F antibody: number analyzed (Participants) | 155 | 158
  Anti-19F antibody | 2.25 [2.02 to 2.50] | 2.10 [1.87 to 2.37]
  Anti-23F antibody: number analyzed (Participants) | 156 | 157
  Anti-23F antibody | 0.94 [0.80 to 1.10] | 0.80 [0.67 to 0.94]
Statistical Analysis 1: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 1 concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 1 is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; GMC adjusted for BS sub cohorts;97.5% CI for adjusted GMC ratio (Ancova Model: adjustment for BS sub cohorts-pooled variance); Adjusted GMC ratio = 1.18, 97.5% CI 2-sided [0.95 to 1.47] — To be able to conclude independently on primary objectives of Epoch 001(Rotarix & Prevnar13 post dose 3)& Epoch 002(Havrix & Prevnar13 post dose 4),Bonferroni correction is used to test these primary objectives(1.25% 1sided for Epoch 001 & Epoch 002)
Statistical Analysis 2: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 3 concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 3 is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; GMC adjusted for BS subcohorts;97.5% CI for the adjusted GMC ratio(Ancova model:adjustment for BS subcohorts-pooled variance); Adjusted GMC ratio = 1.15, 97.5% CI 2-sided [0.93 to 1.42] — To be able to conclude independently on primary objectives of Epoch 001(Rotarix & Prevnar13 post dose 3)& Epoch 002(Havrix&Prevnar13 post dose 4),a Bonferroni correction is used to test these primary objectives(1.25% 1sided for Epoch 001 & Epoch 002)
Statistical Analysis 3: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 4 concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 4 is to be≥ 0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.08, 97.5% CI 2-sided [0.90 to 1.31] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 5 concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 5 is to be ≥ 0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.18, 97.5% CI 2-sided [0.95 to 1.47] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 6A concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 6A is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.29, 97.5% CI 2-sided [1.03 to 1.63] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 6B concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 6B is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.17, 97.5% CI 2-sided [0.88 to 1.55] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 7F concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 7F is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.11, 97.5% CI 2-sided [0.91 to 1.34] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 9V concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 9V is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.25, 97.5% CI 2-sided [1.00 to 1.55] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 14 concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 14 is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.16, 97.5% CI 2-sided [0.90 to 1.50] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 18C concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 18C is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.24, 97.5% CI 2-sided [1.01 to 1.52] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 11: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 19A concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 19A is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.16, 97.5% CI 2-sided [0.94 to 1.43] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 12: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 19F concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 19F is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.07, 97.5% CI 2-sided [0.89 to 1.29] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 13: Comparison: HibCY Group vs PedHIB Group; GMC ratio between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 23F concentrations one month after the third dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 23F is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 3, analysis 2]; Adjusted GMC ratio = 1.18, 97.5% CI 2-sided [0.91 to 1.53] — [estimate comment as in outcome 3, analysis 2]

4. Primary Outcome: Percentage of Subjects With Anti-Hepatitis A (Anti-Havrix) Antibody Concentrations ≥ 15mIU/mL
Description: Percentage of subjects with Anti-Havrix (Anti-HAV) antibody concentrations was assessed. The cut-off value is ≥15 mIU/mL.
  Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.As per an hierarchical procedure, the primary objective about Anti-PRP will first need to be met to be able to conclude on any other primary objective, and within each subsequent arm, the first primary objective will have to be reached to conclude on the second primary objective of that Epoch
Time Frame: 1 month post-dose 2 of Havrix (Month 17-20)
Population: The analysis was performed on the Havrix ATP cohort for analysis of immunogenicity which include all evaluable subjects who received two doses of Havrix vaccine and for whom immunogenicity results were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 129 | 124
Percentage of subjects | 100 [97.2 to 100] | 100 [97.1 to 100]
Statistical Analysis 1: Comparison: HibCY Group vs PedHIB Group; Difference between HibCY and PedHIB groups in percentage of subjects with anti-HAV concentrations equal to or above the cut-off value of 15 mIU/mL one month after the second Havrix dose; Test type: Non-Inferiority — Lower limit of the two-sided standardized asymptotic 97.5% CI on the difference (HibCY group minus the PedHIB group) in the percentage of subjects with anti-HAV concentrations ≥15 mIU/mL is to be≥-10% (clinical limit for non-inferiority); Group difference in proportions; Difference in percentage of subjects = 0.00, 97.5% CI 2-sided [-3.76 to 3.91] — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: Anti-S. Pneumoniae GMCs
Description: as for outcome 3
Time Frame: 1 month post-dose 4 of Prevnar 13 (Month 11-14)
Population: The analysis was performed on the Forth dose ATP cohort for analysis of immunogenicity, which included all evaluable subjects who have received four doses of Prevnar 13 vaccine and for whom immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 216 | 205
µg/mL
  Anti-1 antibody | 2.00 [1.78 to 2.25] | 1.60 [1.43 to 1.79]
  Anti-3 antibody: number analyzed (Participants) | 169 | 167
  Anti-3 antibody | 0.52 [0.46 to 0.58] | 0.51 [0.44 to 0.59]
  Anti-4 antibody | 1.36 [1.23 to 1.50] | 1.24 [1.10 to 1.39]
  Anti-5 antibody: number analyzed (Participants) | 215 | 205
  Anti-5 antibody | 2.36 [2.10 to 2.64] | 2.23 [1.97 to 2.52]
  Anti-6A antibody | 6.80 [6.10 to 7.57] | 5.63 [5.05 to 6.26]
  Anti-6B antibody: number analyzed (Participants) | 215 | 205
  Anti-6B antibody | 5.57 [4.97 to 6.24] | 4.94 [4.40 to 5.55]
  Anti-7F antibody | 4.16 [3.76 to 4.61] | 3.81 [3.45 to 4.21]
  Anti-9V antibody: number analyzed (Participants) | 215 | 205
  Anti-9V antibody | 1.38 [1.25 to 1.53] | 1.24 [1.11 to 1.39]
  Anti-14 antibody | 7.14 [6.32 to 8.07] | 6.13 [5.48 to 6.86]
  Anti-18C antibody: number analyzed (Participants) | 216 | 204
  Anti-18C antibody | 1.62 [1.46 to 1.80] | 1.42 [1.28 to 1.57]
  Anti-19A antibody: number analyzed (Participants) | 216 | 204
  Anti-19A antibody | 5.47 [4.87 to 6.14] | 5.03 [4.47 to 5.64]
  Anti-19F antibody: number analyzed (Participants) | 215 | 205
  Anti-19F antibody | 6.23 [5.61 to 6.92] | 5.54 [4.97 to 6.18]
  Anti-23F antibody | 3.28 [2.90 to 3.71] | 2.68 [2.37 to 3.05]
Statistical Analysis 1: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 1 concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 1 is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; GMC adjusted for BS sub cohorts;97.5% CI for adjusted GMC ratio(Ancova model:adjustment for BS sub cohorts-pooled variance); Adjusted GMC ratio = 1.25, 97.5% CI 2-sided [1.04 to 1.51] — To be able to conclude independently on primary objectives of Epoch 001 & Epoch 002, a Bonferroni correction is used to test these primary objectives(1.25% one-sided for Epoch 001 and Epoch 002)
Statistical Analysis 2: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 3 concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 3 is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.01, 97.5% CI 2-sided [0.83 to 1.24] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 4 concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 4 is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.10, 97.5% CI 2-sided [0.92 to 1.31] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 5 concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 5 is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.06, 97.5% CI 2-sided [0.87 to 1.28] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 6A concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 6A is to be≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.21, 97.5% CI 2-sided [1.01 to 1.44] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 6B concentrations one month after the fourth dose; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 6]; ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.13, 97.5% CI 2-sided [0.94 to 1.36] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 7F concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 7F is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.09, 97.5% CI 2-sided [0.93 to 1.29] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 9V concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 9V is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.12, 97.5% CI 2-sided [0.94 to 1.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 14 concentrations one month after the fourth dose; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 9]; ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.16, 97.5% CI 2-sided [0.96 to 1.41] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 18C concentrations one month after the fourth dose; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.14, 97.5% CI 2-sided [0.97 to 1.35] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 19A concentrations one month after the fourth dose; Test type: Non-Inferiority — Lower limit of the two-sided 97.5% CI on the GMC ratio (HibCY group over PedHIB group) for antibodies to S. pneumoniae serotype 19A is to be ≥0.5 (clinical limit for non-inferiority); ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.09, 97.5% CI 2-sided [0.90 to 1.31] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 19F concentrations one month after the fourth dose; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 12]; ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.12, 97.5% CI 2-sided [0.95 to 1.34] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: HibCY Group vs PedHIB Group; GMC ratios between HibCY and PedHIB groups for antibodies to S. pneumoniae serotype 23F concentrations one month after the fourth dose; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 13]; ANCOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 1.22, 97.5% CI 2-sided [1.00 to 1.50] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Subjects With Anti-PRP Antibody Concentrations ≥0.15 µg/mL.
Description: The cut-off value for this assay was 0.15 µg/mL. Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 2 months post-dose 2 [PedHib Group only (Month 4)], 1 month post-dose 3 (Month 5 for HibCY group and Months 11-14 for PedHib Group) and 1 month post-dose 4 [HibCY Group only (Month 11-14)]
Population: The analysis was performed on the First three doses ATP cohort for analysis of immunogenicity (for Month 4 and Month 5) and the Fourth doses ATP cohort for analysis of immunogenicity (for Months 11-14) which included all evaluable subjects for whom immunogenicity results were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 223 | 218
Percentage of subjects
  Month 4: number analyzed (Participants) | 0 | 165
  Month 4 |  | 98.8 [95.7 to 99.9]
  Month 5: number analyzed (Participants) | 167 | 0
  Month 5 | 99.4 [96.7 to 100] |
  Month 11-14 | 99.6 [97.5 to 100] | 100 [98.3 to 100]

7. Secondary Outcome: Anti-PRP GMCs≥ 0.15 µg/mL.
Description: Anti-PRP antibody concentrations were assessed by Enzyme-Linked-Immunosorbent-Assay (ELISA), tabulated as Geometric Mean Concentrations (GMCs) and expressed in micrograms per mililiter (µg/mL).The cut-off value for this assay was 0.15 µg/mL.
  Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 2 months post-dose 2 [PedHib Group only (Month 4)], 1 month post-dose 3 (Month 5 for HibCY group and Month 11-14 for PedHib Group) and 1 month post-dose 4 [HibCY Group only (Month 11-14)]
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 223 | 218
µg/mL
  Month 4: number analyzed (Participants) | 0 | 165
  Month 4 |  | 11.053 [8.740 to 13.979]
  Month 5: number analyzed (Participants) | 167 | 0
  Month 5 | 8.414 [7.070 to 10.014] |
  Month 11-14 | 28.090 [24.012 to 32.862] | 20.869 [17.799 to 24.468]

8. Secondary Outcome: Percentage of Subjects With Anti-PRP Antibody Concentrations ≥1.0 µg/mL
Description: The cut-off value for this assay was 1.0 µg/mL. Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 2 months post-dose 2 [PedHib group only (Month 4)] and 1 month postdose 3 [HibCY group only (Month 5)].
Population: The analysis was performed on the First three doses ATP cohort for analysis of immunogenicity (for Month 4 and Month 5) which included all evaluable subjects for whom immunogenicity results were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- HibCY Group: Subjects received 4 doses of Hib-MenCY-TT vaccine at Day 0, Month 2, Month 4 and Month 10-13 , 3 doses of Pediarix® vaccine at Day 0, Month 2 and Month 4, 2 doses of Rotarix® vaccine at Day 0 and Month 2, 4 doses of Prevnar 13® vaccine at Day 0 and Month 2, Month 4 and Month 10-13 and 2 doses of Havrix® vaccine at Month 10-13 and Month 16-19.
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 167 | 165
Percentage of subjects
  Month 4: number analyzed (Participants) | 0 | 165
  Month 4 |  | 91.5 [86.2 to 95.3]
  Month 5: number analyzed (Participants) | 167 | 0
  Month 5 | 94.0 [89.3 to 97.1] |

9. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Assay to N. Meningitidis Serogroup C (hSBA-MenC) and N. Meningitidis Serogroup Y (hSBA-MenY) Antibody Titers ≥1:8, ≥1:16, ≥1:32.
Description: The cut off values are dilutions of 1:8, 1:16 and 1:32. Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 1 month post-dose 3 (Month 5) and 1 month post-dose 4 (Month 11-14).
Population: The analysis was performed on the First three doses ATP cohort for analysis of immunogenicity (for Month 5) and the Fourth doses ATP cohort for analysis of immunogenicity (for Months11-14) which included all evaluable subjects for whom immunogenicity results were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 215 | 187
Percentage of subjects
  hSBA-MenC, Month 5, ≥ 8: number analyzed (Participants) | 144 | 141
  hSBA-MenC, Month 5, ≥ 8 | 100 [97.5 to 100] | 1.4 [0.2 to 5.0]
  hSBA-MenC, Month 5, ≥ 16: number analyzed (Participants) | 144 | 141
  hSBA-MenC, Month 5, ≥ 16 | 100 [97.5 to 100] | 1.4 [0.2 to 5.0]
  hSBA-MenC, Month 5, ≥ 32: number analyzed (Participants) | 144 | 141
  hSBA-MenC, Month 5, ≥ 32 | 99.3 [96.2 to 100] | 0.7 [0.0 to 3.9]
  hSBA-MenY, Month 5, ≥ 8: number analyzed (Participants) | 130 | 150
  hSBA-MenY, Month 5, ≥ 8 | 97.7 [93.4 to 99.5] | 100 [97.6 to 100]
  hSBA-MenY, Month 5, ≥ 16: number analyzed (Participants) | 130 | 150
  hSBA-MenY, Month 5, ≥ 16 | 97.7 [93.4 to 99.5] | 100 [97.6 to 100]
  hSBA-MenY, Month 5, ≥ 32: number analyzed (Participants) | 130 | 150
  hSBA-MenY, Month 5, ≥ 32 | 97.7 [93.4 to 99.5] | 100 [97.6 to 100]
  hSBA-MenC, Month 11-14, ≥ 8: number analyzed (Participants) | 215 | 168
  hSBA-MenC, Month 11-14, ≥ 8 | 99.1 [96.7 to 99.9] | 0.6 [0.0 to 3.3]
  hSBA-MenC, Month 11-14, ≥ 16: number analyzed (Participants) | 215 | 168
  hSBA-MenC, Month 11-14, ≥ 16 | 98.6 [96.0 to 99.7] | 0.6 [0.0 to 3.3]
  hSBA-MenC, Month 11-14, ≥ 32: number analyzed (Participants) | 215 | 168
  hSBA-MenC, Month 11-14, ≥ 32 | 98.1 [95.3 to 99.5] | 0.0 [0.0 to 2.2]
  hSBA-MenY, Month 11-14, ≥ 8: number analyzed (Participants) | 198 | 187
  hSBA-MenY, Month 11-14, ≥ 8 | 98.5 [95.6 to 99.7] | 100 [98.0 to 100]
  hSBA-MenY, Month 11-14, ≥ 16: number analyzed (Participants) | 198 | 187
  hSBA-MenY, Month 11-14, ≥ 16 | 98.5 [95.6 to 99.7] | 100 [98.0 to 100]
  hSBA-MenY, Month 11-14, ≥ 32: number analyzed (Participants) | 198 | 187
  hSBA-MenY, Month 11-14, ≥ 32 | 98.5 [95.6 to 99.7] | 100 [98.0 to 100]

10. Secondary Outcome: Geometric Mean Titres (GMTs) of Human Complement Serum Bactericidal Assay to N. Meningitidis Serogroup C (hSBA-MenC) and to hSBA-MenY
Description: The cut-off values are dilutions of 1:8, 1:16 and 1:32. Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 1 month post-dose 3 (Month 5) and 1 month post-dose 4 (Month 11-14).
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 215 | 187
Titres
  hSBA-MenC, Month 5: number analyzed (Participants) | 144 | 141
  hSBA-MenC, Month 5 | 807.3 [659.2 to 988.6] | 2.1 [2.0 to 2.3]
  hSBA-MenY, Month 5: number analyzed (Participants) | 130 | 150
  hSBA-MenY, Month 5 | 510.9 [405.7 to 643.3] | 550.2 [474.4 to 638.1]
  hSBA-MenC, Month 11-14: number analyzed (Participants) | 215 | 168
  hSBA-MenC, Month 11-14 | 2566.2 [2046.3 to 3218.1] | 2.0 [2.0 to 2.1]
  hSBA-MenY, Month 11-14: number analyzed (Participants) | 198 | 187
  hSBA-MenY, Month 11-14 | 2761.4 [2274.2 to 3353.1] | 2728.2 [2412.7 to 3085.0]

11. Secondary Outcome: Percentage of Subjects With Anti-rotavirus IgA Antibody Concentrations ≥ 20 Units (U)/mL
Description: The cut-off value is 20 Units (U)/mL Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 2 month post-dose 2 of Rotarix (Month 4)
Population: The analysis was performed on the Rota ATP cohort for analysis of immunogenicity which included all vaccinated subjects for whom data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 155 | 161
Percentage of subjects | 81.3 [74.2 to 87.1] | 80.1 [73.1 to 86.0]

12. Secondary Outcome: Percentage of Subjects With Anti-HAV Antibodies ≥ 15 mIU/mL
Description: The cut-off value is 15 mIU/mL. Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups.
Time Frame: 1 month post-dose 1 of Havrix (Month 11-14)
Population: The analysis was performed on the Fourth dose ATP cohort for analysis of immunogenicity, which included all vaccinated subjects for whom data are available.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 182 | 168
percentage of subjects | 85.2 [79.2 to 90.0] | 89.3 [83.6 to 93.5]

13. Secondary Outcome: Anti-HAV GMCs ≥ 15 mIU/mL
Description: as for outcome 12
Time Frame: 1 month post-dose 1 of HAV (M11-14).
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 182 | 168
mIU/mL | 44.8 [38.3 to 52.5] | 47.3 [40.9 to 54.8]

14. Secondary Outcome: GMCs for Anti-HAV Antibodies ≥15mIU/mL.
Description: as for outcome 12
Time Frame: 1 month post-dose 2 of HAV (Month 17-20).
Population: This analysis was performed on Havrix ATP cohort for analysis of immunogenicity which included all evaluable subjects who have received the first and second dose of Havrix and for whom assay results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 129 | 124
mIU/mL | 1590.7 [1312.7 to 1927.5] | 1390.6 [1147.8 to 1684.6]

15. Secondary Outcome: Percentage of Subjects With S. Pneumoniae Antibody Concentrations ≥ 0.15 µg/mL, ≥ 0.26 µg/mL and ≥ 0.35 µg/mL for Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F
Description: The cut-off values are 0.15, 0.26, 0.35 µg/mL. Analysis of Immunogenicity is performed on blood sample (BS) sub-cohorts.Assignment to a BS sub-cohort depends on the date of enrolment of the subject: BS sub-cohort for the first 200 , for the next 200 subjects or for the last 200 subjects. Within each BS sub-cohort subjects have been randomized 1:1 to either HibCY or PedHIB groups
Time Frame: 1 month post-dose 3 (Month 5) and 1 month post-dose 4 (Month 11-14)
Population: This analysis was perfomed on First three doses ATP for analysis of immunogenicity and on the Fourth dose ATP cohort for analysis of immunogenicity which included all evaluable subjects for whom data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 216 | 205
Percentage of subjects
  Anti-1 antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-1 antibody, Month 5, ≥ 0.15 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Anti-1 antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-1 antibody, Month 5, ≥ 0.26 | 98.1 [94.5 to 99.6] | 98.7 [95.5 to 99.8]
  Anti-1 antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-1 antibody, Month 5, ≥ 0.35 | 96.8 [92.7 to 99.0] | 93.7 [88.7 to 96.9]
  Anti-3 antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 149 | 150
  Anti-3 antibody, Month 5, ≥ 0.15 | 96.6 [92.3 to 98.9] | 94.0 [88.9 to 97.2]
  Anti-3 antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 149 | 150
  Anti-3 antibody, Month 5, ≥ 0.26 | 84.6 [77.7 to 90.0] | 78.7 [71.2 to 84.9]
  Anti-3 antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 149 | 150
  Anti-3 antibody, Month 5, ≥ 0.35 | 69.8 [61.7 to 77.0] | 69.3 [61.3 to 76.6]
  Anti-4 antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-4 antibody, Month 5, ≥ 0.15 | 98.7 [95.4 to 99.8] | 98.1 [94.6 to 99.6]
  Anti-4 antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-4 antibody, Month 5, ≥ 0.26 | 96.8 [92.7 to 99.0] | 91.8 [86.3 to 95.5]
  Anti-4 antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-4 antibody, Month 5, ≥ 0.35 | 91.0 [85.4 to 95.0] | 84.8 [78.2 to 90.0]
  Anti-5 antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-5 antibody, Month 5, ≥ 0.15 | 97.4 [93.6 to 99.3] | 96.8 [92.8 to 99.0]
  Anti-5 antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-5 antibody, Month 5, ≥ 0.26 | 93.6 [88.5 to 96.9] | 86.7 [80.4 to 91.6]
  Anti-5 antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-5 antibody, Month 5, ≥ 0.35 | 91.0 [85.4 to 95.0] | 80.4 [73.3 to 86.3]
  Anti-6A antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-6A antibody, Month 5, ≥ 0.15 | 100 [97.7 to 100] | 98.7 [95.5 to 99.8]
  Anti-6A antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-6A antibody, Month 5, ≥ 0.26 | 98.7 [95.4 to 99.8] | 94.3 [89.5 to 97.4]
  Anti-6A antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-6A antibody, Month 5, ≥ 0.35 | 98.1 [94.5 to 99.6] | 91.8 [86.3 to 95.5]
  Anti-6B antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 154 | 158
  Anti-6B antibody, Month 5, ≥ 0.15 | 95.5 [90.9 to 98.2] | 93.7 [88.7 to 96.9]
  Anti-6B antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 154 | 158
  Anti-6B antibody, Month 5, ≥ 0.26 | 90.9 [85.2 to 94.9] | 86.1 [79.7 to 91.1]
  Anti-6B antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 154 | 158
  Anti-6B antibody, Month 5, ≥ 0.35 | 83.8 [77.0 to 89.2] | 80.4 [73.3 to 86.3]
  Anti-7F antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-7F antibody, Month 5, ≥ 0.15 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Anti-7F antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-7F antibody, Month 5, ≥ 0.26 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Anti-7F antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-7F antibody, Month 5, ≥ 0.35 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Anti-9V antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 157
  Anti-9V antibody, Month 5, ≥ 0.15 | 99.4 [96.5 to 100] | 94.9 [90.2 to 97.8]
  Anti-9V antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 157
  Anti-9V antibody, Month 5, ≥ 0.26 | 92.9 [87.7 to 96.4] | 86.6 [80.3 to 91.5]
  Anti-9V antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 157
  Anti-9V antibody, Month 5, ≥ 0.35 | 83.3 [76.5 to 88.8] | 76.4 [69.0 to 82.8]
  Anti-14 antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 156
  Anti-14 antibody, Month 5, ≥ 0.15 | 100 [97.7 to 100] | 99.4 [96.5 to 100]
  Anti-14 antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 156
  Anti-14 antibody, Month 5, ≥ 0.26 | 100 [97.7 to 100] | 98.1 [94.5 to 99.6]
  Anti-14 antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 156
  Anti-14 antibody, Month 5, ≥ 0.35 | 99.4 [96.5 to 100] | 97.4 [93.6 to 99.3]
  Anti-18C antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-18C antibody, Month 5, ≥ 0.15 | 100 [97.7 to 100] | 98.1 [94.6 to 99.6]
  Anti-18C antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-18C antibody, Month 5, ≥ 0.26 | 96.8 [92.7 to 99.0] | 91.1 [85.6 to 95.1]
  Anti-18C antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-18C antibody, Month 5, ≥ 0.35 | 87.2 [80.9 to 92.0] | 82.3 [75.4 to 87.9]
  Anti-19A antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 158
  Anti-19A antibody, Month 5, ≥ 0.15 | 100 [97.7 to 100] | 98.1 [94.6 to 99.6]
  Anti-19A antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 158
  Anti-19A antibody, Month 5, ≥ 0.26 | 99.4 [96.5 to 100] | 93.0 [87.9 to 96.5]
  Anti-19A antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 158
  Anti-19A antibody, Month 5, ≥ 0.35 | 97.4 [93.6 to 99.3] | 90.5 [84.8 to 94.6]
  Anti-19F antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 155 | 158
  Anti-19F antibody, Month 5, ≥ 0.15 | 100 [97.6 to 100] | 100 [97.7 to 100]
  Anti-19F antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 155 | 158
  Anti-19F antibody, Month 5, ≥ 0.26 | 100 [97.6 to 100] | 100 [97.7 to 100]
  Anti-19F antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 155 | 158
  Anti-19F antibody, Month 5, ≥ 0.35 | 98.7 [95.4 to 99.8] | 100 [97.7 to 100]
  Anti-23F antibody, Month 5, ≥ 0.15: number analyzed (Participants) | 156 | 157
  Anti-23F antibody, Month 5, ≥ 0.15 | 96.8 [92.7 to 99.0] | 96.2 [91.9 to 98.6]
  Anti-23F antibody, Month 5, ≥ 0.26: number analyzed (Participants) | 156 | 157
  Anti-23F antibody, Month 5, ≥ 0.26 | 91.7 [86.2 to 95.5] | 84.1 [77.4 to 89.4]
  Anti-23F antibody, Month 5, ≥ 0.35: number analyzed (Participants) | 156 | 157
  Anti-23F antibody, Month 5, ≥ 0.35 | 83.3 [76.5 to 88.8] | 77.1 [69.7 to 83.4]
  Anti-1 antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-1 antibody, Month 11-14, ≥ 0.26 | 99.5 [97.4 to 100] | 99.5 [97.3 to 100]
  Anti-1 antibody, Month 11-14, ≥0.35 | 97.7 [94.7 to 99.2] | 97.1 [93.7 to 98.9]
  Anti-3 antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 169 | 167
  Anti-3 antibody, Month 11-14, ≥ 0.15 | 97.0 [93.2 to 99.0] | 94.0 [89.3 to 97.1]
  Anti-3 antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 169 | 167
  Anti-3 antibody, Month 11-14, ≥ 0.26 | 85.2 [78.9 to 90.2] | 81.4 [74.7 to 87.0]
  Anti-3 antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 169 | 167
  Anti-3 antibody, Month 11-14, ≥0.35 | 71.6 [64.2 to 78.3] | 69.5 [61.9 to 76.3]
  Anti-4 antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 98.5 [95.8 to 99.7]
  Anti-4 antibody, Month 11-14, ≥ 0.26 | 98.6 [96.0 to 99.7] | 97.1 [93.7 to 98.9]
  Anti-4 antibody, Month 11-14, ≥0.35 | 97.7 [94.7 to 99.2] | 94.1 [90.0 to 96.9]
  Anti-5 antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 215 | 205
  Anti-5 antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-5 antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 215 | 205
  Anti-5 antibody, Month 11-14, ≥ 0.26 | 99.5 [97.4 to 100] | 99.5 [97.3 to 100]
  Anti-5 antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 215 | 205
  Anti-5 antibody, Month 11-14, ≥0.35 | 99.1 [96.7 to 99.9] | 98.0 [95.1 to 99.5]
  Anti-6A antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-6A antibody, Month 11-14, ≥ 0.26 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-6A antibody, Month 11-14, ≥0.35 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-6B antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 215 | 205
  Anti-6B antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-6B antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 215 | 205
  Anti-6B antibody, Month 11-14, ≥ 0.26 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-6B antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 215 | 205
  Anti-6B antibody, Month 11-14, ≥0.35 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-7F antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-7F antibody, Month 11-14, ≥ 0.26 | 100 [98.3 to 100] | 99.5 [97.3 to 100]
  Anti-7F antibody, Month 11-14, ≥0.35 | 100 [98.3 to 100] | 99.5 [97.3 to 100]
  Anti-9V antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 215 | 205
  Anti-9V antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 99.0 [96.5 to 99.9]
  Anti-9V antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 215 | 205
  Anti-9V antibody, Month 11-14, ≥ 0.26 | 99.1 [96.7 to 99.9] | 98.5 [95.8 to 99.7]
  Anti-9V antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 215 | 205
  Anti-9V antibody, Month 11-14, ≥0.35 | 97.7 [94.7 to 99.2] | 96.6 [93.1 to 98.6]
  Anti-14 antibody, Month 11-14, ≥ 0.15 | 99.5 [97.4 to 100] | 100 [98.2 to 100]
  Anti-14 antibody, Month 11-14, ≥ 0.26 | 99.5 [97.4 to 100] | 100 [98.2 to 100]
  Anti-14 antibody, Month 11-14, ≥0.35 | 99.5 [97.4 to 100] | 100 [98.2 to 100]
  Anti-18C antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 216 | 204
  Anti-18C antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-18C antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 216 | 204
  Anti-18C antibody, Month 11-14, ≥ 0.26 | 99.5 [97.4 to 100] | 99.0 [96.5 to 99.9]
  Anti-18C antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 216 | 204
  Anti-18C antibody, Month 11-14, ≥0.35 | 98.6 [96.0 to 99.7] | 97.5 [94.4 to 99.2]
  Anti-19A antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 216 | 204
  Anti-19A antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-19A antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 216 | 204
  Anti-19A antibody, Month 11-14, ≥ 0.26 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-19A antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 216 | 204
  Anti-19A antibody, Month 11-14, ≥0.35 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-19F antibody, Month 11-14, ≥ 0.15: number analyzed (Participants) | 215 | 205
  Anti-19F antibody, Month 11-14, ≥ 0.15 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-19F antibody, Month 11-14, ≥ 0.26: number analyzed (Participants) | 215 | 205
  Anti-19F antibody, Month 11-14, ≥ 0.26 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-19F antibody, Month 11-14, ≥0.35: number analyzed (Participants) | 215 | 205
  Anti-19F antibody, Month 11-14, ≥0.35 | 100 [98.3 to 100] | 100 [98.2 to 100]
  Anti-23F antibody, Month 11-14, ≥ 0.15 | 99.5 [97.4 to 100] | 100 [98.2 to 100]
  Anti-23F antibody, Month 11-14, ≥ 0.26 | 99.5 [97.4 to 100] | 100 [98.2 to 100]
  Anti-23F antibody, Month 11-14, ≥0.35 | 98.1 [95.3 to 99.5] | 100 [98.2 to 100]

16. Secondary Outcome: Percentage of Subjects Reporting Any Solicited Local Adverse Events (AE).
Description: Solicited local adverse events include pain, redness and swelling at injection site.
Time Frame: 4 days (Day 0 to Day 3) after all vaccines post-primary and post-fourth dose
Population: This analysis was performed on First three doses Total Vaccinated cohort and on the Fourth dose total vaccinated cohort which included all evaluable subjects who received atleast one dose of any of the study vaccines:Hib-MenCY-TT, Pediarix, Prevnar 13, Rotarix, PedvaxHIB or Havrix, and with the vaccine administration documented.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 285 | 291
Percentage of subjects
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 1 | 44.2 [38.4 to 50.2] | 61.2 [55.3 to 66.8]
  Pain, Pediarix, Dose 1 | 50.5 [44.6 to 56.5] | 57.4 [51.5 to 63.1]
  Pain, Prevnar 13, Dose 1 | 46.3 [40.4 to 52.3] | 58.8 [52.9 to 64.5]
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 2: number analyzed (Participants) | 272 | 278
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 2 | 45.6 [39.6 to 51.7] | 56.8 [50.8 to 62.7]
  Pain, Pediarix, Dose 2: number analyzed (Participants) | 272 | 278
  Pain, Pediarix, Dose 2 | 45.2 [39.2 to 51.3] | 55.8 [49.7 to 61.7]
  Pain, Prevnar 13, Dose 2: number analyzed (Participants) | 272 | 277
  Pain, Prevnar 13, Dose 2 | 44.5 [38.5 to 50.6] | 56.0 [49.9 to 61.9]
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 3: number analyzed (Participants) | 260 | 0
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 3 | 38.8 [32.9 to 45.1] |
  Pain, Pediarix, Dose 3: number analyzed (Participants) | 262 | 264
  Pain, Pediarix, Dose 3 | 42.7 [36.7 to 49.0] | 50.8 [44.6 to 56.9]
  Pain, Prevnar 13, Dose 3: number analyzed (Participants) | 262 | 264
  Pain, Prevnar 13, Dose 3 | 39.7 [33.7 to 45.9] | 47.7 [41.6 to 53.9]
  Pain,Havrix , Dose 4: number analyzed (Participants) | 241 | 242
  Pain,Havrix , Dose 4 | 44.8 [38.4 to 51.3] | 50.0 [43.5 to 56.5]
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 4: number analyzed (Participants) | 241 | 242
  Pain, Hib-MenCY-TT/PedvaxHIB, Dose 4 | 42.3 [36.0 to 48.8] | 56.2 [49.7 to 62.5]
  Pain, Prevnar 13, Dose 4: number analyzed (Participants) | 241 | 242
  Pain, Prevnar 13, Dose 4 | 41.5 [35.2 to 48.0] | 46.7 [40.3 to 53.2]
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 1: number analyzed (Participants) | 284 | 291
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 1 | 21.1 [16.5 to 26.3] | 35.4 [29.9 to 41.2]
  Redness, Pediarix, Dose 1: number analyzed (Participants) | 284 | 291
  Redness, Pediarix, Dose 1 | 27.1 [22.0 to 32.7] | 25.1 [20.2 to 30.5]
  Redness, Prevnar 13, Dose 1: number analyzed (Participants) | 284 | 291
  Redness, Prevnar 13, Dose 1 | 23.6 [18.8 to 29.0] | 24.4 [19.6 to 29.8]
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 2: number analyzed (Participants) | 271 | 278
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 2 | 30.3 [24.8 to 36.1] | 41.4 [35.5 to 47.4]
  Redness, Pediarix, Dose 2: number analyzed (Participants) | 271 | 278
  Redness, Pediarix, Dose 2 | 33.9 [28.3 to 39.9] | 43.2 [37.3 to 49.2]
  Redness, Prevnar 13, Dose 2: number analyzed (Participants) | 271 | 277
  Redness, Prevnar 13, Dose 2 | 30.6 [25.2 to 36.5] | 41.2 [35.3 to 47.2]
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 3: number analyzed (Participants) | 260 | 0
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 3 | 31.5 [25.9 to 37.6] |
  Redness, Pediarix, Dose 3: number analyzed (Participants) | 262 | 264
  Redness, Pediarix, Dose 3 | 38.2 [32.3 to 44.3] | 50.4 [44.2 to 56.6]
  Redness, Prevnar 13, Dose 3: number analyzed (Participants) | 262 | 264
  Redness, Prevnar 13, Dose 3 | 36.3 [30.4 to 42.4] | 45.8 [39.7 to 52.1]
  Redness,Havrix , Dose 4: number analyzed (Participants) | 241 | 242
  Redness,Havrix , Dose 4 | 38.6 [32.4 to 45.1] | 43.8 [37.5 to 50.3]
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 4: number analyzed (Participants) | 241 | 242
  Redness, Hib-MenCY-TT/PedvaxHIB, Dose 4 | 38.6 [32.4 to 45.1] | 50.8 [44.3 to 57.3]
  Redness, Prevnar 13, Dose 4: number analyzed (Participants) | 241 | 242
  Redness, Prevnar 13, Dose 4 | 41.1 [34.8 to 47.6] | 44.6 [38.3 to 51.1]
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 1: number analyzed (Participants) | 284 | 291
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 1 | 11.3 [7.8 to 15.5] | 22.0 [17.4 to 27.2]
  Swelling, Pediarix, Dose 1: number analyzed (Participants) | 284 | 291
  Swelling, Pediarix, Dose 1 | 18.7 [14.3 to 23.7] | 16.2 [12.1 to 20.9]
  Swelling, Prevnar 13, Dose 1: number analyzed (Participants) | 284 | 291
  Swelling, Prevnar 13, Dose 1 | 14.8 [10.9 to 19.5] | 16.2 [12.1 to 20.9]
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 2: number analyzed (Participants) | 271 | 278
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 2 | 18.5 [14.0 to 23.6] | 30.6 [25.2 to 36.4]
  Swelling, Pediarix, Dose 2: number analyzed (Participants) | 271 | 278
  Swelling, Pediarix, Dose 2 | 22.1 [17.3 to 27.6] | 36.3 [30.7 to 42.3]
  Swelling, Prevnar 13, Dose 2: number analyzed (Participants) | 271 | 277
  Swelling, Prevnar 13, Dose 2 | 22.5 [17.7 to 28.0] | 28.9 [23.6 to 34.6]
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 3: number analyzed (Participants) | 260 | 0
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 3 | 19.2 [14.6 to 24.6] |
  Swelling, Pediarix, Dose 3: number analyzed (Participants) | 262 | 264
  Swelling, Pediarix, Dose 3 | 29.4 [23.9 to 35.3] | 37.9 [32.0 to 44.0]
  Swelling, Prevnar 13, Dose 3: number analyzed (Participants) | 262 | 264
  Swelling, Prevnar 13, Dose 3 | 24.4 [19.3 to 30.1] | 31.4 [25.9 to 37.4]
  Swelling,Havrix , Dose 4: number analyzed (Participants) | 241 | 242
  Swelling,Havrix , Dose 4 | 25.3 [19.9 to 31.3] | 26.0 [20.6 to 32.0]
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 4: number analyzed (Participants) | 241 | 242
  Swelling, Hib-MenCY-TT/PedvaxHIB, Dose 4 | 22.8 [17.7 to 28.6] | 34.3 [28.3 to 40.6]
  Swelling, Prevnar 13, Dose 4: number analyzed (Participants) | 241 | 242
  Swelling, Prevnar 13, Dose 4 | 26.1 [20.7 to 32.2] | 27.7 [22.1 to 33.8]

17. Secondary Outcome: Percentage of Subjects Reporting Any Solicited General AEs.
Description: Solicited general AEs include fever [defined as temperature ≥38.0 degrees Celsius (°C) by any method], drowsiness, irritability/fussiness and loss of appetite.
Time Frame: 4 days (Day 0 to Day 3) after all vaccines post-primary and post-fourth dose.
Population: The analysis was performed on First three doses Total Vaccinated cohort and on the Fourth dose Total Vaccinated cohort which included all evaluable subjects who received atleast one dose of any of the study vaccines:Hib-MenCY-TT, Pediarix, Prevnar 13, Rotarix, PedvaxHIB or Havrix, and with the vaccine administration documented.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 285 | 291
Percentage of subjects
  Any Temperature (°C), Dose 1 | 11.2 [7.8 to 15.5] | 20.6 [16.1 to 25.7]
  Any Temperature (°C), Dose 2: number analyzed (Participants) | 273 | 279
  Any Temperature (°C), Dose 2 | 19.4 [14.9 to 24.6] | 29.0 [23.8 to 34.7]
  Any Temperature (°C), Dose 3: number analyzed (Participants) | 262 | 265
  Any Temperature (°C), Dose 3 | 16.4 [12.1 to 21.5] | 17.0 [12.7 to 22.1]
  Any Temperature (°C), Dose 4: number analyzed (Participants) | 242 | 241
  Any Temperature (°C), Dose 4 | 8.7 [5.5 to 13.0] | 10.4 [6.8 to 14.9]
  Irritability / Fussiness, Dose 1 | 71.2 [65.6 to 76.4] | 81.8 [76.9 to 86.0]
  Irritability / Fussiness, Dose 2: number analyzed (Participants) | 273 | 278
  Irritability / Fussiness, Dose 2 | 70.0 [64.1 to 75.3] | 83.5 [78.6 to 87.6]
  Irritability / Fussiness, Dose 3: number analyzed (Participants) | 262 | 265
  Irritability / Fussiness, Dose 3 | 66.0 [59.9 to 71.7] | 69.4 [63.5 to 74.9]
  Irritability / Fussiness, Dose 4: number analyzed (Participants) | 241 | 241
  Irritability / Fussiness, Dose 4 | 66.0 [59.6 to 71.9] | 74.3 [68.3 to 79.7]
  Loss Of Appetite, Dose 1 | 31.6 [26.2 to 37.3] | 42.3 [36.5 to 48.2]
  Loss Of Appetite, Dose 2: number analyzed (Participants) | 273 | 278
  Loss Of Appetite, Dose 2 | 29.7 [24.3 to 35.5] | 31.7 [26.2 to 37.5]
  Loss Of Appetite, Dose 3: number analyzed (Participants) | 262 | 265
  Loss Of Appetite, Dose 3 | 29.8 [24.3 to 35.7] | 28.7 [23.3 to 34.5]
  Loss Of Appetite, Dose 4: number analyzed (Participants) | 241 | 241
  Loss Of Appetite, Dose 4 | 33.2 [27.3 to 39.5] | 39.8 [33.6 to 46.3]
  Drowsiness, Dose 1 | 64.9 [59.1 to 70.4] | 70.1 [64.5 to 75.3]
  Drowsiness, Dose 2: number analyzed (Participants) | 273 | 278
  Drowsiness, Dose 2 | 54.2 [48.1 to 60.2] | 65.1 [59.2 to 70.7]
  Drowsiness, Dose 3: number analyzed (Participants) | 262 | 265
  Drowsiness, Dose 3 | 48.9 [42.7 to 55.1] | 52.5 [46.3 to 58.6]
  Drowsiness, Dose 4: number analyzed (Participants) | 241 | 241
  Drowsiness, Dose 4 | 44.0 [37.6 to 50.5] | 48.5 [42.1 to 55.0]

18. Secondary Outcome: Percentage of Subjects Reporting Any Unsolicited AEs.
Description: Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms were reported as an unsolicited adverse event.
Time Frame: During 31 days (Day 0 to Day 30) after all vaccines post-primary (Dose 1-3) and post-fourth dose (Dose 4)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 297 | 303
Percentage of subjects
  Dose 1-3 | 60.6 [54.8 to 66.2] | 56.4 [50.6 to 62.1]
  Dose 4: number analyzed (Participants) | 248 | 250
  Dose 4 | 39.9 [33.8 to 46.3] | 42.0 [35.8 to 48.4]

19. Secondary Outcome: Percentage of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Month 17-20)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HibCY Group | PedHIB Group
Number analyzed (Participants) | 297 | 303
Percentage of subjects | 2.7 [1.2 to 5.2] | 3.6 [1.8 to 6.4]

ADVERSE EVENTS:
Time Frame: Solicited adverse events - Day 0-Day 4 Unsolicited Adverse events - Day 0- Day 31 after all vaccines post-primary and post-fourth dose. SAEs - day 0 to study end (Month 17-20)
Arm/Group | HibCY Group | PedHIB Group
All-Cause Mortality (participants affected / at risk) | 1/297 | 0/303
Serious Adverse Events (participants affected / at risk) | 8/297 | 11/303
Other Adverse Events (participants affected / at risk) | 282/297 | 291/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HibCY Group (N=297) | PedHIB Group (N=303)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Kawasaki's disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HibCY Group (N=297) | PedHIB Group (N=303)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Administration site haemorrhage (General disorders) | 1 (1) | 0 (0)
Administration site rash (General disorders) | 0 (0) | 1 (1)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Body height below normal (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Bronchiolitis (Infections and infestations) | 13 (13) | 9 (9)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 3 (3) | 4 (4)
Candida nappy rash (Infections and infestations) | 1 (1) | 4 (4)
Cardiac murmur (Investigations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Communication disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 11 (11) | 16 (17)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (13) | 9 (11)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 31 (32)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 10 (10)
Cyanosis (Cardiac disorders) | 0 (0) | 2 (2)
Dacryocystitis (Infections and infestations) | 1 (1) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 2 (2) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 177 (331) | 200 (384)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 (11) | 15 (15)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 14 (15) | 12 (13)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 26 (31) | 18 (20)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 6 (9) | 5 (9)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (8)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema infectiosum (Infections and infestations) | 1 (1) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (6) | 3 (3)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Fontanelle depressed (Nervous system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 2 (2) | 3 (3)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Frenulum breve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 4 (4)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 7 (7) | 12 (12)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 13 (13)
Genital labial adhesions (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 3 (3) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Herpangina (Infections and infestations) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 5 (5) | 3 (3)
Injection site erythema (General disorders) | 189 (442) | 211 (539)
Injection site induration (General disorders) | 2 (2) | 2 (2)
Injection site mass (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 229 (550) | 248 (648)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 147 (322) | 182 (413)
Injection site warmth (General disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 267 (737) | 284 (839)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Language disorder (Nervous system disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Macrocephaly (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 2 (3) | 1 (1)
Motor developmental delay (Nervous system disorders) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1) | 1 (1)
Mycoplasma test positive (Investigations) | 1 (1) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 15 (15)
Nasopharyngitis (Infections and infestations) | 16 (17) | 12 (14)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 2 (2)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 43 (48) | 41 (49)
Otitis media acute (Infections and infestations) | 6 (6) | 5 (6)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Penile adhesion (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 6 (7)
Plagiocephaly (Congenital, familial and genetic disorders) | 6 (6) | 6 (6)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Poor feeding infant (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Positional plagiocephaly (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 124 (184) | 147 (235)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 13 (14)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (12)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 19 (21)
Roseola (Infections and infestations) | 2 (2) | 1 (1)
Screaming (Psychiatric disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Selective eating disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 5 (5) | 2 (2)
Skin candida (Infections and infestations) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 230 (569) | 254 (641)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 13 (13) | 13 (13)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 62 (78) | 35 (40)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Vaccination site induration (General disorders) | 0 (0) | 1 (2)
Vaccination site nodule (General disorders) | 0 (0) | 1 (1)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 8 (8) | 9 (9)
Viral rash (Infections and infestations) | 5 (5) | 4 (5)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 14 (14) | 20 (24)
Vomiting projectile (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Weight (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.